CLINICAL TRIAL: NCT02233374
Title: Predicting RadIotherapy ReSponse of Rectal Cancer With MRI and PET
Acronym: PRISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, Professor Andrew Kneebone, Associate Professor Andrew Kneebone, Royal North Shore Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-NSCCRO-P001
Record Dates: First submitted 2014-08-13; First posted 2014-09-08 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Rectal Neoplasms
Keywords: Rectal Cancer; Magnetic Resonance Imaging; Positron Emission Tomography; pathologic complete response; Diffusion-weighted magnetic resonance imaging; Microstructural Imaging; FDG PET
MeSH Terms: conditions — Rectal Neoplasms; Pathologic Complete Response | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Assessing response with MRI + PET. (Experimental): Pre-operative chemo/RT as per standard treatment. Intensity Modulated Radiotherapy (IMRT) / Volumetric Arc Therapy (VMAT) 45Gray/25 fractions with simultaneous integrated Boost of 50Gray/25 fractions + concurrent capecitabine chemotherapy.
  Intervention 1 'Early MRI and PET/CT - 2 weeks after commencing chemo/RT' involves additional Multiparametric MRI + PET/CT 2 weeks into chemo/RT Intervention 2 :\'Late MRI and PET/CT 6 weeks post chemo/RT' involves additional Multiparametric MRI + PET/CT 6 weeks post chemo/RT
  Interventions: Other: Early MRI and PET/CT - 2 weeks after commencing chemo/RT; Other: Late MRI and PET/CT 6 weeks post chemo/RT

INTERVENTIONS:
Other: Early MRI and PET/CT - 2 weeks after commencing chemo/RT — Patients will have an early MRI and PET/CT - 2 weeks after commencing chemo/RT. A limited range PET/CT will look at parameters: SUVmaxm PERCIST, RECIST 1.1, ΔSUV (PET1-2), ΔSUV (early -late), Glycolytic tumour volume (GTV). MRI T2 (1-3mm slice as per NS Radiology protocol and ESGAR guideline) will look at parameters: DWI & ADC value (preferably on a single camera with reproducible ADC value), Local Staging, MRF involvement, EMVI, nodal status, MR volumetry, and desmoplastic reaction.
  Other Names: Imaging
Other: Late MRI and PET/CT 6 weeks post chemo/RT — Patients will have late a MRI and PET/CT 6 weeks post chemo/RT. A whole body PET/CT will look at parameters: SUVmaxm PERCIST, RECIST 1.1, ΔSUV (PET1-2), ΔSUV (early -late), Glycolytic tumour volume (GTV). MRI T2 (1-3mm slice as per NS Radiology protocol and ESGAR guideline) will look at parameters: DWI & ADC value (preferably on a single camera with reproducible ADC value), Local Staging, MRF involvement, EMVI, nodal status, MR volumetry, and desmoplastic reaction.
  Other Names: Imaging

SUMMARY:
The purpose of this study is to investigate if PET/CT and MRI scans performed early in treatment and six weeks after treatment can predict the response of rectal cancer following chemotherapy and radiotherapy. This will help doctors to better tailor treatments for rectal cancer in the future.

DETAILED DESCRIPTION:
Bowel cancer is the second most prevalent cancer in Australia with rectal cancer the most common subgroup, representing 5% of all cancer diagnoses in 2008 [1]. Rectal cancer also accounts for 4.6% of all cancer deaths in New South Wales [1]. All rectal cancer that is T3/4 or node positive on pre-operative assessment should be considered for pre-operative therapy, which has been shown to significantly improve local control compared to postoperative chemoradiation. [2]. Pre-operative chemoradiation is standard pre-operative treatment at the Northern Sydney Cancer Centre with approximately 40 patients/year receiving this treatment. Surgery is normally performed 6-8 weeks following chemoradiation.

One of the unique opportunities with rectal cancer is that histopathological analysis of the resected specimen gives an accurate assessment of the response of the tumour to pre-operative chemoradiation. Those tumours having a pathologic complete response (pCR) are known to have an excellent long-term outcome.

Data from the department of Radiation Oncology at Northern Sydney Cancer Centre demonstrates that only 17% of patients experience a pCR, which is in keeping with other series [4]. In this study of 48 patients, 38% showed evidence of tumour shrinkage 2 weeks into treatment as demonstrated on a Cone Beam CT scan taken during radiotherapy. 44% of these patients demonstrated a pCR following surgery. In the remaining 62%, none of these patients had a pCR. This confirms the principle that early response during radiation based only on gross tumour shrinkage can be a powerful predictor of subsequent response.

Assessing response during Cone Beam CT is very subjective and not possible on all patients. Furthermore it may be possible to better predict those likely to have a complete response with alternate imaging modalities. There is emerging data that functional and microstructural imaging modalities can also be used to predict and assess treatment response prior to, during and following the delivery of pre-operative chemoradiation for locally advanced rectal cancer [5].

Diffusion-weighted magnetic resonance imaging (DWI) is a microstructural imaging technique that characterizes tissue based on differences in the movement of water molecules. These differences can be quantified using the apparent diffusion coefficient (ADC). The ADC has been shown to differentiate post-treatment inflammation and necrosis from recurrent or persistent tumoural tissue in rectal cancer with high specificity [6]. Pre-treatment ADC assessment with DWI has a sensitivity of 100% and specificity of 86% for detection of pCR (p=0.003) whilst treatment induced changes in ADC (measured at week 2 chemoradiation) have a sensitivity and specificity of 100% for predicting pCR (p=0.0006) [5]. Prediction of response should be improved further with the use of PET imaging. A staging 18F-FDG (18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose ) PET/CT has been demonstrated to provide new findings compared to contrast-enhanced CT of the thorax/abdomen/pelvis resulting in a change in the stage of disease and alteration of treatment strategy in 14% of patients [7]. F-FDG PET/CT can be more predictive of histological response and outcome than anatomic imaging alone [8]. Whilst PET Response Criteria in Solid Tumors (PERCIST) has not been shown to have predictive power on the response to neoadjuvant therapy, PET Residual Disease in Solid Tumor (PREDIST) criteria has been shown to correlate to pCR (p = 0.004) [9].

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* T3/4 or node positive rectal cancer
* Suitable for pre-operative chemo-irradiation and surgical resection
* No contraindication to MRI (pacemaker, severe claustrophobia)
* Gross visible disease on MRI
* No contraindications to PET/CT
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Karnofsky Performance Status > 70%)
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* - Previous radiotherapy to pelvis
* Unable/unwilling to have MRI
* Unable/unwilling to have PET/CT
* Pregnancy, lactation or inadequate contraception
* Known allergic reaction to FDG PET contrast
* Pacemaker or implanted defibrillator
* Patients with a history of psychological illness or condition such as to interfere with the patient's ability to understand requirements of the study.
* Unwilling or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Predictive value of PET/CT and MRI 2 weeks into chemo-irradiation for developing a pathologic complete response at surgery. | 2 years
  Predictive value of PET/CT and MRI 2 weeks into chemo-irradiation for developing a pathologic complete response at surgery (Grade 0 - no viable cancer cells seen in the resection specimen).
  The standard grading system employed by pathologists at Royal North Shore Hospital will be used to measure tumour regression. This is the system recommended by the RCPA synoptic report for colorectal cancer, based on Ryan R, Gibbons D, Hyland JMP, et al. Pathological response following long-course neoadjuvant chemoradiotherapy for locally advanced rectal cancer. Histopathology 2005; 47:141-6.

SECONDARY OUTCOMES:
Feasibility of conducting additional PET and MRI scans at 6 weeks post-treatment. | 2 years
  This will be assessed in terms of whether PET and MR imaging approximately 6 weeks after chemo-irradiation adds any additional predictive value to imaging performed 2 weeks into treatment.
Utility of adding PET scan to the baseline staging of patients | 2 years
  This will be measured by whether PET 2 weeks into treatment (combined with already utilised MRI) can independently predict the likelihood of a pathological complete response at surgery.
Pathologic response according to Tumour Regression Grade (TRG) | 2.5 years
  A scoring system will be developed based on the degree of response from the PET and MRI scan at 2 weeks incorporating tumour shrinkage (PET and MR), reduction in SUV (PET) and reduction in diffusion (MR) that can best predict the "responders" and "non-responders".
Impact of pCR rates on long term disease control | 5 years
  Measured in terms of loco-regional or distant recurrence by 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kneebone, MBBS, Principal Investigator — Royal North Shore Hospital
Locations (1):
- Northern Sydney Cancer Centre, Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No